CLINICAL TRIAL: NCT02435199
Title: A Double-blind, Placebo-controlled, Randomized Trial to Determine the Safety and Efficacy of EMA401 in Patients With Painful Diabetic Neuropathy
Brief Title: Clinical Trial Designed to Determine the Safety and Efficacy of EMA401 in Patients With Painful Diabetic Neuropathy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Spinifex Pharmaceuticals Pty Ltd (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMA401-011
Record Dates: First submitted 2015-04-24; First posted 2015-05-06 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — EMA400

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMA401 600mg (Experimental): 2 X 150mg BID
  Interventions: Drug: EMA401 600mg
- Placebo (Placebo Comparator): Placebo to match, 2 capsules BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EMA401 600mg
  Arms: EMA401 600mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study consists of two periods, the Screening Period (~3 weeks) and Treatment Period (12 weeks).

Eligibility for the study will be determined by Screening tests, physical examination/medical history, and fulfilment of eligibility criteria including assessment of pain completed during the Screening Period. Potential participants will be required to provide written informed consent prior to any study-specific Screening procedures being performed.

Following Screening assessments, patients will be randomized to receive either EMA401 300 mg BID or placebo.

Patient study visits during the Treatment Period are at the end of baseline/randomization visit, and end of Weeks 3, 6, 9, and 12, for assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type I or Type II diabetes mellitus with painful, distal, symmetrical, sensory-motor neuropathy attributed to diabetes, of at least six months duration.
* Be assessed as suffering from moderate to severe pain across the Screening Period. The assessment of moderate and severe pain will be made using an algorithm proprietary to Spinifex. The investigator/site staff will be informed immediately as to whether the patient is eligible or ineligible on the ePRO website based on the patient entering all relevant pain scores in the eDiary device.
* Women of child bearing potential (WOCBP), must have a negative urine pregnancy test at the Screening visit (Visit 1) and within 72 hours prior to administration of IP.

Exclusion Criteria:

* Patients taking any topical treatment for their PDN at the time of Screening Visit 2 will be excluded, including lidocaine plaster, capsaicin patch, and any other topical preparations of these or any other topical medications (e.g., aspirin, Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) for their PDN.
* Have a blood pressure reading, after resting for at least five minutes, outside a systolic blood pressure range of 84 - 151 mmHg or a diastolic blood pressure > 95 mmHg. If the blood pressure is outside of the range, a repeat measurement can be taken after the patient has rested. The repeat measurement should be used as the screening value.
* Have serum aspartate transaminase (AST), or alanine transaminase (ALT) levels > 1.5 x the upper limit of normal or have total bilirubin concentrations > 1.5 x the upper limit of normal at Screening (Visit 1).
* Have hemoglobin A1c > 11 %.
* Known history of, or positive laboratory results for hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) infection as defined by being seropositive for hepatitis B surface antigen (HBsAg), HCV antibodies or HIV antibodies respectively.
* Have undergone neurolytic or neurosurgical therapy or use a neurostimulating device for PDN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of EMA401 compared to placebo in patients with painful diabetic neuropathy (PDN), as assessed by the difference in the weekly mean of the 24 hour average pain score, using an 11-point Numeric Rating Scale (NRS). | Change from Baseline to Week 12

SECONDARY OUTCOMES:
The effect of EMA401 compared to placebo on the BPI-SF interference total score. | Change from Baseline to Week 12
The effect of EMA401 compared to placebo on the weekly mean of the 24 hour worst NRS pain score. | Change from Baseline to Week 12
The effect of EMA401 compared to placebo, on the Patient Global Impression of Change (PGIC). | Change from Baseline to Week 12
The effect of EMA401 compared to placebo on the Brief Pain Inventory-Short Form (BPI-SF) average pain score. | Change from Baseline to Week 12
The proportion of EMA401 patients achieving a ≥ 30% and a ≥ 50% reduction in weekly mean 24 hour average pain score compared to placebo (i.e., responder rates). | Change from Baseline to Week 12
The effect of EMA401 compared to placebo on the Neuropathic Pain Symptom Inventory (NPSI). | Change from Baseline to Week 12
The effect of EMA401 compared to placebo on the Insomnia Severity Index (ISI). | Change from Baseline to Week 12
The safety and tolerability of EMA401 in patients with PDN as measured by number and severity of adverse events. | Change from Baseline to Week 12